CLINICAL TRIAL: NCT05596682
Title: Prospective Multicenter Clinical Study on the Visual and Refractive Outcomes and Safety Outcomes Following Implantation of an AddOn Intraocular Lens in Previously Pseudophakic Eyes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medicontur Medical Engineering Ltd (Industry)
Collaborators: Medevise Consulting (Unknown)
Responsible Party: Sponsor
Other Study IDs: MC_AddOn_multi_2020
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Presbyopia; Refractive Errors; Residual Astigmatism
MeSH Terms: conditions — Presbyopia; Refractive Errors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: supplementary intraocular lenses — Implantation of supplementary intraocular lenses into the ciliary sulcus in previously pseudophakic eyes.
  Other Names: 1stQ AddOn

SUMMARY:
The purpose of this prospective multicenter clinical study is to evaluate the visual and refractive outcomes and safety outcomes following bilateral implantation of trifocal and/or trifocal toric 1stQ AddOn (Medicontur) intraocular lenses (IOLs) to correct residual refractive errors, astigmatism, and presbyopia in previously pseudophakic eyes.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read and sign the Informed Consent form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Adult males or females above 18 years of age.
4. No other ocular co -morbidity (i.e. no history of ocular surface disease, severe dry eye, glaucoma, retinal or macular pathology)
5. Pseudophakia.
6. Uncomplicated cataract surgery or clear lens extraction followed by an uneventful recovery period of at least 3-months.
7. Stable primary IOL located in the capsular bag.
8. Anterior chamber depth (ACD) of at least 2.8 mm (measured from corneal endothelium to the anterior surface of the primary IOL in the capsular bag with an optical biometer [Lenstar, IOL Master]).
9. Subjects with residual refractive error that is suitable for correction with a secondary add-on IOL.
10. Subjects, who have stable post-operative refraction at month two following uncomplicated primary lens surgery.
11. Subjects with myopia of not more than 6.0 diopters.
12. Subjects with monocular corrected distance visual acuity (CDVA) of Snellen 6/7.5 (20/25; LogMAR=0.1, decimal=0.80) or better.
13. Subjects with a preoperative pharmacologically dilated pupil diameter of 6.5 mm or more.

Exclusion Criteria:

1. Currently pregnant or lactating.
2. Prisoners or young offenders in custody
3. Adults lacking capacity to consent for themselves
4. Phakic or aphakic status.
5. Narrow angle, i.e. < Schaefer grade 2
6. Pseudophakic patients with malpositioned, subluxated or unstable capsular fixated intraocular lens.
7. Patients with a multifocal capsular bag fixated IOL.
8. Inability to achieve secure placement in the designated location e.g. due to absence of a secure peripheral anterior capsule, absence of intact zonules, or irregular anatomy of the ciliary sulcus.
9. Active ocular diseases (chronic severe uveitis, proliferative diabetic retinopathy, chronic glaucoma not responsive to medication, iris atrophy, severe zonulopathy, pigment dispersion syndrome).
10. Corneal abnormalities such as Unstable Keratoconus, irregular astigmatism.
11. Existing ocular conditions such as age-related macular degeneration (AMD) and other progressive retinal degenerations.
12. Any previous ocular co-morbidity including pseudoexfoliation, zonular weakness, pseudophakodonesis, complicated cataract surgery, narrow angle glaucoma or macular pathology, congenital eye abnormality, microphthalmia.
13. Any eye disease in which postoperative visual acuity is not expected to be better than 0.5 decimal (e.g. amblyopia, nystagmus, retinitis pigmentosa, aniridia, eccentric pupil)
14. Subjects with pathological pupil reactions.
15. Subjects with untreated posterior capsule opacification (PCO), which results in at least 1-line decrease in visual acuity and/or in loss of contrast sensitivity (CS).
16. Any systemic disease (e.g., Sjögren's syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with visual function and/or participation in the study.
17. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with visual function.
18. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with visual function and/or participation in the study.
19. Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.)
20. Any greater than Grade 2 slit lamp findings (e.g., oedema, corneal neovascularisation, corneal staining, tarsal abnormalities, conjunctival injection, corneal decompensation) or any other ocular abnormality that may contraindicate the implantation of the supplementary IOL.
21. Any history or signs of a corneal inflammatory event, or any other ocular abnormality
22. Participation in any intraocular lens, contact lens or lens care product clinical trial within 30 days prior to study enrollment.
23. Employee, relative or friends of employees of any ophthalmic company, or investigational clinic (e.g., Investigator, Coordinator, Technician)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pseudophakic subjects after uncomplicated implantation of a monofocal intraocular lens (IOL) in the capsular bag who have elected to undergo a secondary add-on IOL procedure to correct presbyopia and/or the residual refractive and/or cylindric error after primary lens implantation
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Distance Corrected Near Visual Acuity (DCNVA) | 6 months
  Monocular and binocular DCNVA changes at 6 months after IOLs implantation in comparison to Baseline.

SECONDARY OUTCOMES:
Distance Corrected Near Visual Acuity (DCNVA) | 12 months
  Monocular and binocular DCNVA changes after IOLs implantation in comparison to Baseline.
Uncorrected Near Visual Acuity (UNVA) | 12 months
  Monocular and binocular UNVA after IOLs implantation
Uncorrected Intermediate Visual Acuity (UIVA) | 12 months
  Monocular and binocular UIVA after IOLs implantation
Distance Corrected Intermediate Visual Acuity (DCIVA) | 12 months
  Monocular and binocular DCIVA after IOLs implantation
Uncorrected Distance Visual Acuity (UDVA) | 12 months
  Monocular and binocular UDVA after IOLs implantation
Corrected Distance Visual Acuity (CDVA) | 12 months
  Monocular and binocular CDVA after IOLs implantation

CONTACTS AND LOCATIONS:
Overall Officials: Prof Sathish Srinivasan, Principal Investigator — Ayrshire Eye Clinic
Locations (4):
- Medipolis Antwerp Private Clinic, Antwerp, Belgium
- Institut Ophtalmologique de l'Ouest Jules Verne, Nantes, France
- Hospital Vithas Almería, Almería, Spain
- Ayrshire Eye Clinic, Ayr, Scotland, United Kingdom